CLINICAL TRIAL: NCT02797366
Title: Proton Radiotherapy for Primary Central Nervous System Tumours in Adults - a Prospective Swedish Multicentre Study
Brief Title: Proton Radiotherapy for Primary Central Nervous System Tumours in Adults
Acronym: PRO-CNS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); University Hospital, Umeå (Other); Region Örebro County (Other); University Hospital, Linkoeping (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-CNS
Record Dates: First submitted 2016-05-18; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Central Nervous System Tumour; Arteriovenous Malformation
MeSH Terms: conditions — Arteriovenous Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton radiotherapy (Other): Proton radiation therapy daily (Monday through Friday) for 4-8 weeks. This is a single arm study.
  Interventions: Radiation: Proton radiotherapy

INTERVENTIONS:
Radiation: Proton radiotherapy

SUMMARY:
Open label, multi-centre prospective study. Adult patients with primary central nervous system tumours fulfilling the inclusion criteria according to the study protocol. The study consists of 2 sequential cohorts evaluated consecutively for the feasibility, safety and toxicity, as well as long-term survival data, when using spot scanning proton beam therapy.

DETAILED DESCRIPTION:
Open label, multi-centre prospective phase II study. Adult patients with primary central nervous system tumours full-filling the inclusion criteria according to the study protocol. The study consists of 2 sequential cohorts evaluated for the feasibility, safety and toxicity, as well as long-term survival data, when using proton beam therapy.

* Part I: To assess the feasibility of using pencil beam scanning and evaluating the treatment safety in all aspects, and to assess acute toxicity in a smaller cohort of CNS patients. All toxicity data, QoL and survival data will also be included in the part II cohort.
* Part II: The second part of the trial consists of all CNS patients that are referred to the Skandion Clinic after the safety data from the first part has been evaluated by the study steering committee.

ELIGIBILITY:
Inclusion criteria:

* The patient must be at least 18 years old
* World Health Organization (WHO)/ Eastern Cooperative OncologyGroup (ECOG) performance status 0-2, Karnofsky score ≥60.
* The patient must be able to understand the information about the treatment and give a written informed consent to participate in the trial.
* Adequate follow-up study must be possible; this will exclude a patient who is uncooperative.
* Must have a life expectancy of at least 3 years based on age and co-morbidities as well as diagnosis. For patients considered for re-irradiation the life expectancy must be estimated to minimum 6 months.
* Must have a pathology proven CNS tumour or if not possible, the radiology findings must be evaluated at a multi-disciplinary conference at a university hospital.
* Women of reproductive potential must agree to use an effective method of contraception during therapy such as an intrauterine device or condom. Pregnancy IS not an ineligibility criteria if radiotherapy is indicated and can-not be postponed.
* Prior CNS radiotherapy is not an ineligibility criteria but re-irradiated patients will be included in a subgroup evaluated separately.

Patients discussed at multidisciplinary conferences at one of the seven university hospitals in Sweden and found candidates for radiotherapy and one of following diagnoses:

* Anaplastic glioma grade III with Loss of Heterozygosity (LOH) 1p/19q and isocitrate dehydrogenase-1 (IDH-1) mutation
* Arteriovenous malformations (AVMs)
* Chordomas and chondrosarcomas
* Craniopharyngiomas
* Ependymomas
* Intracranial germ cell tumours
* Low grade gliomas - grade I-II
* Medulloblastoma, Primitive neuroectodermal tumour (PNET)
* Meningiomas
* Neurocytoma
* Other grade I-II primary CNS tumour according to WHO classification
* Pituitary adenomas
* Schwannomas
* Spinal tumours
* Whenever craniospinal irradiation (CSI) is indicated
* Whenever re-irradiation of CNS is considered

Exclusion criteria:

* Concomitant or previous malignancies. Exceptions are adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, or in situ carcinoma of the cervix uteri with a follow-up time of at least 3 years, or other previous malignancy with a disease-free interval of at least 5 years.
* Not able to understand information or manage tests according to study protocol. If necessary, only authorized interpreters may be used to assist in the translation.
* Psychiatric or addictive disorders or other medical conditions that, in the opinions of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Acute adverse events | 3 months
Long-term adverse events | 10-15 years
  This study specifically includes longitudinal follow-up to assess the incidence of neurotoxicity including cognitive dysfunction, as well as the incidence of secondary malignant neoplasms at 10 and 15 years following radiotherapy.

SECONDARY OUTCOMES:
Local and regional tumour control | 15 years
  Including overall survival
Pattern of failure | 15 years
  Pattern of failure on MRI will be compared with patients getting conventional radiotherapy.
Quality of life | 5 years
  Quality of Life (QoL) data will be evaluated using validated questionnaires from the European Organization for Research and Treatment of Cancer (EORTC): EORTC-QLQ-C30 is a multidimensional, cancer-specific QoL questionnaire developed for repeated assessments in clinical trials, and validated in various cancer populations. The Brain Cancer Module (EORTC-QLQ-BN20) includes 20 questions focusing on neurological symptoms and EuroQoL (EQ-5D) may additional also be used in the study.
Normal tissue sparing and normal tissue complication | 15 years
  Normal tissue complication probability (NTCP) models will be used to evaluate the reduction in normal tissue complications in dose planning studies comparing proton radiotherapy vs. 3D-Conformal Radiotherapy (CRT), Intensity Modulated Radiotherapy (IMRT)/Volumetric Modulated Arc Therapy (VMAT)/Helical Tomotherapy (HTT).

CONTACTS AND LOCATIONS:
Overall Officials: Petra Witt Nystrom, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (6):
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Linkoeping University Hospital, Linköping
  - Orebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Umea University Hospital, Umeå
  - Uppsala University Hospital, Uppsala